CLINICAL TRIAL: NCT06812065
Title: Rrandomized Controlled Clinical Trial Named Mild Local Hyperthermia and Hydrogen Peroxide Treat Multiple Warts by Targeting a Single Lesion.
Brief Title: Randomized Controlled Clinical Trial of Hyperthermia and Hydrogen Peroxide 3% in the Treatment of Cutaneous Warts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH20210930
Record Dates: First submitted 2022-01-05; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Warts
Keywords: hyperthermia; Warts; Hydrogen Peroxide
MeSH Terms: conditions — Warts; Hyperthermia | interventions — Hydrogen Peroxide; Solutions

STUDY DESIGN:
Masking Description: Masking Description:
  * Participants blinded to treatment allocation through:
    1. Identical-appearing placebo devices with sham light emission
    2. Opaque containers for topical solutions (H2O2 vs saline)
    3. Separate treatment rooms per study arm
  * Outcome assessors blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Local Hyperthermia at 44℃ (Experimental): As an experimental arm.
  Interventions: Device: Local Hyperthermia at 44℃
- Local 3%H2O2 treatment (Experimental): As an experimental arm
  Interventions: Drug: Hydrogen Peroxide 3 % Topical Solution
- 3%H2O2 for 1 hour, then local hyperthermia at 44℃ for 30 minutes (Experimental): Undergo the hyperthermia treatment of the Local Hyperthermia Group and the dressing treatment of the 3% Hydrogen Peroxide Group. Apply the 3% hydrogen peroxide dressing 1 hour before each hyperthermia session.
  Local Hyperthermia treats the target warts(largest and most severe warts), while medication addresses all warts.
  Interventions: Drug: Hydrogen Peroxide 3 % Topical Solution; Device: Local Hyperthermia at 44℃

INTERVENTIONS:
Drug: Hydrogen Peroxide 3 % Topical Solution — Dressing: Like the Local Hyperthermia Group, use a cotton ball soaked in 3% hydrogen peroxide.
  Irradiation: For seven sessions in three weeks, use simulated infrared light (without heat) with the same frequency as the Local Hyperthermia Group.
  Local Hyperthermia treats the target warts(largest and most severe warts), while medication addresses all warts.
  Arms: 3%H2O2 for 1 hour, then local hyperthermia at 44℃ for 30 minutes; Local 3%H2O2 treatment
Device: Local Hyperthermia at 44℃ — (Patent No: ZL 200820231952.4, Model: YY-WRY-V01, Liaoning Yanyang Medical Instrument Co., Ltd., China) An infrared hyperthermia device was used to apply local hyperthermia at 44°C to the largest wart. The device includes a heating source, an infrared temperature monitor, an adjusting arm, a control circuit for temperature stabilization, and a display. It uses a tungsten-halogen lamp (wavelength: 760-2300 nm, peak at 1200 nm) to maintain the temperature of a 0.5*0.5 cm skin area within ±0.1°C using a non-contact infrared feedback system.Hyperthermia: Conduct 44-degree Celsius, 30-minute sessions. Do it daily for the first 3 days, then 2 sessions every 7 days for 3 weeks, for a total of 7 sessions.
  Dressing: Apply a cotton ball soaked in 0.9% saline to the warts, wrap it with plastic film for 1 hour, and do this once a day for 6 weeks. Local Hyperthermia treats the target warts(largest and most severe warts), while medication addresses all warts.
  Arms: 3%H2O2 for 1 hour, then local hyperthermia at 44℃ for 30 minutes; Local Hyperthermia at 44℃

SUMMARY:
Hyperthermia treatment (hyperthermia) refers to treating diseases with temperature (39-45 ° C) beyond normal body temperature,. It has been reported that local warming at 44 ° C is able to effectively mobilize the body's immunity and clear HPV infected lesions, such as condyloma acuminatum and verruca vulgaris, etc.

Hydrogen peroxide (H2O2) is a commonly used disinfectant for skin debridement. It has been reported that high concentration of H2O2 (45% H2O2) is effective in the treatment of warts vulgaris, however, high concentration of H2O2 will cause more local pain, itching and burning sensation. 3% hydrogen peroxide is commonly used as skin debridement disinfectant.

The purpose of the study is to evaluate the efficacy and safety of 44℃ hyperthermia combined with 3% hydrogen peroxide in treating verruca virus.

DETAILED DESCRIPTION:
Mild local Hyperthermia with a certain temperature range has been successfully used to treat some diseases. The warm treatment is usually "all or nothing". "All" means that all viral warts are removed after "warm" treatment, including rashes in non-treated areas. "Nothing" means that some viral warts do not respond to heat. Therefore, further enhancing the therapeutic effect of warmth and improving the reaction of some patients is the priority. Cellular experimental studies have found that low concentrations of dioxygen can promote the secretion of a keratinocyte series of inflammatory factors induced by warming. A randomized parallel control design was used to compare the efficacy of hyperthermia combined with hydrogen peroxide therapy and single use of hyperthermia and hydrogen peroxide alone in the treatment of viral warts. Primary analysis: Modified ITT (all randomized patients receiving ≥1 treatment).Missing data: Multiple imputation using chained equations (MICE)

.Between-group comparisons: ANOVA with Tukey posthoc test for continuous variables; Chi-square with Bonferroni correction for categorical variables.Survival analysis: Cox proportional hazards model adjusted for baseline lesion size

ELIGIBILITY:
Inclusion criteria: The participants were between 16 and 65 years of age, had a clinical diagnosis of viral warts (including common warts, plantar warts, or condyloma acuminatum), and could understand and sign informed consent.

Exclusion criteria: presented with clinically atypical warts; had immunocompromised status or a history of HIV infection; received HPV vaccination within the past 6 months; used immunomodulators, immunosuppressants, or systemic corticosteroids within defined timeframes (4 months and 1 month, respectively); underwent local therapies (e.g., laser, cryotherapy, retinoids) on or near warts within protocol-specified intervals; had a history of cutaneous malignancies or current precancerous lesions; exhibited active dermatologic/systemic diseases (e.g., psoriasis, eczema) or skin conditions (e.g., sunburn) potentially increasing study risks; or were deemed ineligible by investigators for other medical or logistical reasons.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete clearance rate of warts | 6 months after the first time of treatment.
  The complete clearance rate was defined as the proportion of patients with lesions that completely disappeared within 6 months of completing all treatments.
Time to complete clearance | 6 months after the first time of treatment.
  Median duration from first treatment to complete resolution (days)
Recurrence rate of warts | recurrence was the proportion of patients with reappearance of lesions at previously cleared sites within 6 months after treatment.
  Complete clearance was defined as the proportion of patients with complete disappearance of lesions within 6 months of completion of all treatments, and recurrence was the proportion of patients with recurrence of lesions at the cured lesion site within 6 and 12 months after treatment,

SECONDARY OUTCOMES:
Changes in the size and number of warts at different points in time | At 1 week, 2 weeks, 3 weeks, 4 weeks, 12 weeks, 24 weeks follow-up
  Changes in the size and number of warts at different time points (1 week, 2 weeks, 3 weeks, 4 weeks, 12 weeks, 24 weeks)
Curative effect of different types of warts | followed up at 6 months
  The cure of different types of warts (common warts, plantar warts, condyloma acuminatum) was followed up at 6 months.
Occurrence of adverse events | During treatment and follow-up
  occurrence of adverse events (short - and long-term adverse reactions) (e.g. blisters, erythema, nail changes, ulcers/scars, hyperpigmentation, hypopigmentation, erosion)
Treatment-related pain intensity | During each treatment session (Day 1, 2, 3, 10, 11, 18, 19)
  Pain assessed by Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain)
Patient satisfaction score | At 6-month follow-up
  Self-reported satisfaction on a 5-point Likert scale (0=very dissatisfied, 5=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Study Director — First Hospital of China Medical University
Locations (2):
- China (2):
  - Guo Hao, Shenyang, Liaoning
  - infrared hyperthermia device (Patent No: ZL 200820231952.4, Model: YY-WRY-V01, Liaoning Yanyang Medical Instrument Co., Ltd., China), Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No